CLINICAL TRIAL: NCT00500110
Title: Neoadjuvant Hormonal Ablation, Imatinib Mesylate and Docetaxel Followed by Radical Prostatectomy for High-Risk Localized Prostate Cancer
Brief Title: Hormonal Ablation, Imatinib Mesylate and Docetaxel for Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0112
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Hormonal Ablation; Docetaxel; Imatinib Mesylate; STI571; Gleevec; Taxotere; Goserelin Acetate; Zoladex; Leuprolide; Lupron
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Imatinib Mesylate; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hormonal Ablation, Imatinib + Docetaxel (Experimental): Imatinib Mesylate 600 mg by mouth (PO) daily + Docetaxel 30 mg/m^2 by vein (IV) weekly + Hormonal Ablation (Goserelin Acetate or Leuprolide) injections every other month or every 3 months
  Interventions: Drug: Docetaxel; Drug: Imatinib Mesylate; Drug: Leuprolide; Drug: Goserelin Acetate

INTERVENTIONS:
Drug: Docetaxel — 30 mg/m^2 by vein (IV) Weekly Over 60 Minutes on Days 1, 8, 15, and 22. This will be followed by 2 weeks with no docetaxel.
  Other Names: Taxotere
Drug: Imatinib Mesylate — 600 mg by mouth (PO) Daily x 42 Days.
  Other Names: Gleevec; STI571
Drug: Leuprolide — Hormone injections given every other month or every 3 months, as determined by the doctor.
  Other Names: Lupron
Drug: Goserelin Acetate — Hormone injections given every other month or every 3 months, as determined by the doctor.
  Other Names: Zoladex

SUMMARY:
Primary Objective:

1. To evaluate the pathological complete response rate to neoadjuvant hormonal ablation, Imatinib and Docetaxel (HID) in high-risk localized prostate cancer.

Secondary Objectives:

1. To describe the time to prostate specific antigen (PSA)-progression after neoadjuvant HID and radical prostatectomy in high-risk localized prostate cancer.
2. To correlate pathological response with modulation of the Platelet-Derived Growth Factor Receptor (PDGFR) pathway.

DETAILED DESCRIPTION:
Docetaxel is a drug that was designed to help kill cancer cells. Imatinib mesylate is a drug designed to block cancer cells from growing and dividing. Hormonal treatment with Lupron (leuprolide) or Zoladex (goserelin acetate) is used to lower testosterone levels in the body because prostate cancer cells need testosterone to survive. All patients will have their prostate gland removed after treatment with these drugs.

Before treatment starts, you will be asked questions about your medical history and have a complete physical examination. You will have blood drawn (2 tablespoons) for routine blood tests. You will be asked questions about any medications you are currently taking and have taken in the past. You will have an electrocardiogram (ECG - a test that measures electrical activity of the heart). As part of your standard care for prostate cancer, you will also have a computed tomography (CT) scan (or magnetic resonance imaging ((MRI)) scan) of the abdomen and pelvis along with a bone scan (x-rays of the bones) to see if the prostate cancer has moved to other parts of your body.

For this study, you will receive hormone injections to lower the levels of testosterone in the blood. You will also take imatinib mesylate capsules by mouth and receive treatment with docetaxel by vein to help kill the cancer cells before surgery.

You will receive hormone therapy with either leuprolide or goserelin acetate injections, whichever your doctor feels will give you the most benefit. The hormone injections will be given every other month or every 3 months. During treatment with the hormones, you will also take an anti-androgen drug called Casodex (bicalutamide) by mouth for up to 2 weeks. This drug is being used to help decrease the risks of developing side effects due to the hormone injections (this is the standard of care with hormone treatments). You will take imatinib mesylate capsules every day for 6 weeks starting with the hormone treatments. You will also receive treatment with docetaxel. Docetaxel injections are given by vein over 60 minutes once a week for 4 weeks in a row. This will be followed by 2 weeks with no docetaxel. This 6 week period is considered a course of treatment. You will have up to 3 courses of treatment (18 weeks) with docetaxel. After this treatment is complete, you will have prostate surgery within 4 weeks or when you have fully recovered from treatment.

During treatment, your general health will be monitored and you will have physical exams and blood tests (about 1-2 tablespoons) often to make sure that you are tolerating the treatment safely. If the disease gets worse or you experience intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Before surgery, you will be given a general anesthetic. An incision (cut) will be made in your abdomen (lower stomach area) and your prostate gland and lymph nodes in the pelvis will be removed. Before the procedure, the risks will be explained to you and you will need to sign a separate consent form.

After surgery, you will have check-up visits every 3 months for 1 year, then every 6 months for the rest of your life. At these visits, you will have a physical exam and around 1-2 tablespoons of blood collected for routine lab tests. If your doctor feels it is necessary, you may also have CT scans, bone scans, and/or x-rays. These tests are being done to check if the cancer has come back. If the cancer comes back, you will be removed from the study and your doctor will discuss treatment options with you.

This is an investigational study. The leuprolide or goserelin acetate injections, bicalutamide tablets, imatinib mesylate capsules, and docetaxel injections are all FDA approved and are commercially available. Up to 36 participants will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the prostate that in the opinion of the surgeon is resectable. Ductal adenocarcinoma of the prostate is included.
* All patients must be regarded as low anesthetic risk for radical prostatectomy and confirm their intention to undergo radical prostatectomy at the end of the neoadjuvant therapy.
* All patients must have at least one of the following high-risk features: clinical or pathological T3 disease, or cT2c or PSA>20ng/ml or Gleason 8-10 adenocarcinoma or clinical T2b and PSA>10ng/ml and Gleason 7 adenocarcinoma. The 1992 AJCC staging system will be followed.
* Prior hormonal therapy up to 2 months is permitted; no concurrent ketoconazole is permitted.
* Patients must have adequate bone marrow function defined as an absolute peripheral granulocyte count of >/= 1,500/mm3 and platelet count of >/= 100,000/mm3; adequate hepatic function defined with a total bilirubin of </= 1.5 mg/dl and aspartate aminotransferase (AST or SGOT)/alanine aminotransferase (ALT or SGPT) </= 2 times the upper limits of normal; adequate renal function defined as serum creatinine clearance >/= 40 cc/min (measured or calculated).
* Patients must sign a written informed consent form prior to treatment. All patients must have a surgical and medical oncology consult prior to signing informed consent.

Exclusion Criteria:

* Patients with small cell or sarcomatoid prostate cancers are not eligible.
* Patients with clinical or radiological evidence of metastatic disease
* Prior chemotherapy or experimental agents
* Patients with severe intercurrent infection.
* Patients with The New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina or myocardial infarction (MI) in the last 6 months.
* Contraindications to corticosteroids.
* Uncontrolled severe hypertension, uncontrolled diabetes mellitus, oxygen-dependent lung disease, chronic liver disease or human immunodeficiency virus (HIV) infection.
* Second malignancies (excluding non-melanoma skin cancer) unless disease-free for 3 years.
* Overt psychosis, mental disability or otherwise incompetent to give informed consent or history of non-compliance.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Mathew P, Pisters LL, Wood CG, Papadopoulos JN, Williams DL, Thall PF, Wen S, Horne E, Oborn CJ, Langley R, Fidler IJ, Pettaway CA. Neoadjuvant platelet derived growth factor receptor inhibitor therapy combined with docetaxel and androgen ablation for high risk localized prostate cancer. J Urol. 2009 Jan;181(1):81-7; discussion 87. doi: 10.1016/j.juro.2008.09.006. Epub 2008 Nov 13. PMID 19012911
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at Medical Clinic from 6/13/03 to 11/29/04.
Period: Overall Study
Arm/Group | Hormonal Ablation, Imatinib + Docetaxel
Started | 39
Completed | 36
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Hormonal Ablation, Imatinib + Docetaxel
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Pathological Complete Response
Description: Probability of response, defined as pathological complete remission based on tissue obtained at surgery. Pathological Complete Response (pCR): Patients without gross or microscopic evidence of residual disease at Radical Prostatectomy defined as pCR.
Time Frame: Every 3 months for 1 year, then every 6 months until disease progression or death
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
participants | 0

ADVERSE EVENTS:
Time Frame: 6 years and 3 months
Arm/Group | Hormonal Ablation, Imatinib + Docetaxel
Serious Adverse Events (participants affected / at risk) | 9/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hormonal Ablation, Imatinib + Docetaxel (N=36)
Alanine aminotransferase (Investigations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
acute coronary syndrome (Cardiac disorders) | 1 (1)
fever (General disorders) | 1 (1)
neutrophil count decreased (Investigations) | 1 (1)
thrombosis/embolism (Vascular disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hormonal Ablation, Imatinib + Docetaxel (N=36)
alanine transaminase (Investigations) | 6 (6)
diarrhea (Gastrointestinal disorders) | 4 (8)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
fatigue (General disorders) | 16 (22)
rash (Skin and subcutaneous tissue disorders) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes